CLINICAL TRIAL: NCT03130881
Title: A Phase I Open-label, Multicenter Dose Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics (PK) of PLB1003 in Patients With ALK-positive (ALK+) Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Phase I Study of a Selective ALK Inhibitor PLB1003 in Patients With ALK+ NSCLC.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pearl Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO-PLB1003-20160828
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2017-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLB1003 (Experimental): ALK-positive (ALK+) advanced NSCLC
  Interventions: Drug: PLB1003

INTERVENTIONS:
Drug: PLB1003 — PLB1003 is a capsule and is administered orally.

SUMMARY:
This phase I, first-in-human dose-escalation study was conducted to determine the maximum tolerated dose (MTD), recommended phase II dose (RP2D), dose-limiting toxicities (DLTs), pharmacokinetics (PK) profile, and preliminary antitumor activity of PLB1003.

DETAILED DESCRIPTION:
This is a Phase I, open-label study of PB1003 administered orally to patients with ALK-positive (ALK+) advanced NSCLC. The study includes a Dose-escalation Part (part A) and a Dose Expansion Part (part B). The aim of the part A is to estimate the MTD and to identify the dose limited toxicity(DLT) and the recommended phase II dose (RP2D) for PLB1003 single agent as well as to determine the PK/PD profile. Once response has been observed in certain dose level, then followed by the expansion part to further assess the clinical efficacy and safety of PLB1003 single agent. Aprox 40 patients will be enrolled in PART A, while 12-24 patients for expansion cohort .

PLB1003 is a potent selective ALK inhibitor. PLB1003 acts on cancer by blocking abnormal ALK-mediated signaling, leading to profound tumour growth inhibition in xenografts of non-small cell lung cancer (NSCLC) tumours.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age≥18 years
* Diagnosed with a locally advanced or metastatic non-small cell lung cancer that has progressed despite standard therapy.
* Must have evidence of ALK positivity from the results of molecular pre-screening evaluations
* At least one measurable lesion as per RECIST v1.1
* Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1
* ECOG Performance Status of 0-2

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases that are neurologically unstable or requiring increasing doses of steroids to control, and patients with any CNS deficits.
* Clinically significant, uncontrolled heart diseases. Unstable angina. History of documented congestive heart failure (New York Heart Association functional classification III-IV) .
* Active peptic ulcer disease or gastritis
* Major surgery within 4 weeks prior to starting PLB1003
* Previous anti-cancer and investigational agents within 4 weeks before first dose of PLB1003..
* Pregnant or nursing women
* Involved in other clinical trials < 30 days prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) . | 18 months.
  The maximum tolerated dose (MTD) was defined as the highest dose for a given schedule that was expected to cause DLTs in no more than 33% of patients during the first cycle of treatment.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of PLB1003 and its metabolite. | Day 1-3 PK Run-in period and Day 1-21 Treatment period
  In the study of PK Run-in period, full Pharmacokinetics (PK) profiles of PLB1003 will be obtained following administration of a single oral dose of PLB1003 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics (PK) sampling will include a pre-dose and at the 0.5, 2, 3,4, 6, 9, 10, 12 and 24 hour time points on days 1, 22 of dosing in the first 21-Day cycle of Treatment period, and pre-dose on days 16, 17 and 18 of the first 21-Day cycle of Treatment period.
Maximum plasma concentration observed (Cmax) of PLB1003 and its metabolite. | Day 1-3 PK Run-in period and Day 1-21 Treatment period
  In the study of PK Run-in period, full Pharmacokinetics (PK) profiles of PLB1003 will be obtained following administration of a single oral dose of PLB-1003 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics (PK) sampling will include a pre-dose and at the 0.5, 2, 3,4, 6, 9, 10, 12 and 24 hour time points on days 1, 22 of dosing in the first 21-Day cycle of Treatment period, and pre-dose on days 16, 17 and 18 of the first 21-Day cycle of Treatment period.
Time to Cmax (Tmax) of PLB1003 and its metabolite. | Day 1-3 PK Run-in period and Day 1-21 Treatment period
  In the study of PK Run-in period, full Pharmacokinetics (PK) profiles of PLB1003 will be obtained following administration of a single oral dose of PLB-1003 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics (PK) sampling will include a pre-dose and at the 0.5, 2, 3,4, 6, 9, 10, 12 and 24 hour time points on days 1, 22 of dosing in the first 21-Day cycle of Treatment period, and pre-dose on days 16, 17 and 18 of the first 21-Day cycle of Treatment period.
Preliminary antitumor activity of PLB1003. | 30 months.
  Preliminary antitumor activity of PLB1003 assessed using RECIST1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided